CLINICAL TRIAL: NCT03577587
Title: Effect and Efficacy of the Herbal Galactagogue Silitidil From Milk Thistle in Mothers of Very Preterm Newborns
Brief Title: Efficacy of Herbal Galactagogue Silitidil After Preterm Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Waldkrankenhaus Protestant Hospital, Spandau (Other)
Collaborators: DMK Group (Unknown)
Responsible Party: Principal Investigator, Dr. Hanna Petersen, Head of Institute for Pediatric Nutritional Research at the Waldkrankenhaus Protestant Hospital, Waldkrankenhaus Protestant Hospital, Spandau
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EWK-002
Record Dates: First submitted 2018-01-09; First posted 2018-07-05 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Breast Milk Production; Human Milk Feeding; Hypogalactia; Preterm Infant Nutrition
Keywords: galactagogue; milk thistle; silymarin; Silitidil
MeSH Terms: conditions — Lactation Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verum (Experimental): Silitidil for 21 days
  Interventions: Dietary Supplement: Silitidil for 21 days
- Placebo (Placebo Comparator): Placebo for 21 days
  Interventions: Dietary Supplement: Placebo for 21 days
- Reference group (No Intervention): Non-randomized healthy volunteering mothers after term birth receiving no intervention

INTERVENTIONS:
Dietary Supplement: Silitidil for 21 days — daily ingestion of herbal galactagogue Silitidil over time period of 3 weeks
  Other Names: Silitidil
  Arms: Verum
Dietary Supplement: Placebo for 21 days — daily ingestion of Placebo preparation over time period of 3 weeks
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
After preterm birth mothers often suffer from hypogalactia. Herbal galactogogues can be used in order to increase milk production. In this double-blind, randomized, placebo-controlled clinical trial the effect of Silitidil, an extract from milk thistle, on the postpartal milk production in mothers of very premature newborns is investigated.

DETAILED DESCRIPTION:
Mothers of preterm infants born at a gestational age <= 32 wg are asked to participate in this double-blind, randomized, placebo-controlled interventional trial, where they will receive a preparation of the herbal galactogogue Silitidil or placebo over an intervention period of 3 weeks. The influence of the galactagogue will be investigated by monitoring daily milk production before, during and 1 week after cessation of the intervention. As secondary outcome parameters weight gain, the progress of enteral feeding, and the percentage of human milk feeding on total enteral feeding volumes will be monitored in the newborn infants. Also the breast milk composition (in terms of fatty acids, protein and carbohydrates content) will be investigated and compared between study groups. Saliva and urine probes will be collected at specific time points to survey hormonal reactions during the various phases of lactation and the relation of maternal hormone levels on milk production.

ELIGIBILITY:
Inclusion Criteria:

* mothers after preterm birth <= 32 weeks of gestation
* Age of the newborn 1 - 5 days
* Human milk feeding intended

Exclusion Criteria:

* Ingestion of other galactagogues
* maternal chronical disease requiring therapy (e.g. severe hypothyreosis, preexistent arterial hypertension, Type I or 2 Diabetes, chronic inflammatory bowel disease, severe bronchial asthma, pollinosis)
* medication influencing prolactine levels
* Mastitis at time of enrollment
* mammary tumors or surgery influencing milk production

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Daily milk production (ml/24h) at end of Intervention period | 3 weeks after study initiation
  Daily milk production (ml/24h) according to pumping protocol

SECONDARY OUTCOMES:
Percentual increase in daily milk production | from 0 to 3 weeks after study initiation
  Percentual increase in daily milk production comparing daily milk production (ml/24h) before and at end of intervention
Percentual increase in daily milk production | from 0 to 4 weeks after study initiation
  Percentual increase in daily milk production comparing daily milk production (ml/24h) before and 1 week after intervention
Milk Protein Content during intervention | at 1 week after study initiation
  Protein content in breast milk sample (mg/100ml)
Milk Protein Content at end of intervention | at 3 weeks after study initiation
  Protein content in breast milk sample (mg/100ml)
Milk Protein Content after intervention | at 4 weeks after study initiation
  Protein content in breast milk sample (mg/100ml)
Milk lactose Content during intervention | at 1 week after study initiation
  Lactose content in breast milk sample (mg/100ml)
Milk lactose Content at end of intervention | at 3 weeks after study initiation
  Lactose content in breast milk sample (mg/100ml)
Milk lactose Content after intervention | at 4 weeks after study initiation
  Lactose content in breast milk sample (mg/100ml)
Milk fatty acids Content during intervention | at 1week after study initiation
  Fatty acids content in breast milk sample (mg/100ml)
Milk fatty acids Content at end of intervention | at 3 weeks after study initiation
  Fatty acids content in breast milk sample (mg/100ml)
Milk fatty acids Content after intervention | at 4 weeks after study initiation
  Fatty acids content in breast milk sample (mg/100ml)
Incidence of formula feeding | 4 weeks
  Incidence of (additional) formula feeding at 4 weeks of life
Time point when enteral feeding volumes reach 120 ml/kgbw | 4 weeks
  day of life when enteral feeding volumes of the preterm Infant have reached 120 ml per kg bodyweight
Percentage of human milk feeding | 4 weeks
  Percentage of human milk feeding on total feeding volume of the preterm infant
daily milk production (ml/24h), baseline | at 0, 1 and 2 weeks after study initiation
  Daily milk production (ml/24h) according to pumping protocol
daily milk production (ml/24h), follow-up | 4 weeks after study initiation
  Daily milk production (ml/24h) according to pumping protocol

OTHER OUTCOMES:
Maternal urine oxytocin/creatinin-ratio | 4 weeks
  Maternal urine oxytocin and creatinin levels before and after breast pumping are determined to create oxytocin/creatin-ratio
Maternal Urine prolactin/creatinin-ratio | 4 weeks
  Maternal urine prolactin and creatinin levels before and after breast pumping are determined to create prolactin/creatin-ratio
Maternal alpha-Amylase level in saliva | 4 weeks
  Maternal alpha-amylase levels before and after breast pumping are determined in saliva samples
Maternal cortisol level in saliva | 4 weeks
  Maternal cortisol levels before and after breast pumping are determined in saliva samples
Incidence of mastitis | 4 weeks
  Incidence of clinical mastitis during intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Frank Jochum, MD, Study Director — Head of Paediatric Department
Locations (1):
- Evangelic Waldkrankenhaus Spandau, Paul Gerhardt Diakonie, Berlin-Spandau, Germany

IPD SHARING:
Plan to Share IPD: No